CLINICAL TRIAL: NCT05883020
Title: Effect of Radial Shock Wave Therapy on Calf Muscle Tone, ROM, Gross Motor Scale, Plantar Surface and Quality of Life in Patients With Cerebral Palsy: Randomized Controlled Trial
Brief Title: Effect of Radial Shockwave on Calf Muscle Spasticity in Patients With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hail (Other)
Responsible Party: Principal Investigator, Hisham Mohamed Hussein, principal investigator, University of Hail
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: H-2023-150
Record Dates: First submitted 2023-03-17; First posted 2023-05-31 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Cerebral Palsy
Keywords: radial shockwave therapy; muscle tone; ROM; gross motor scale; quality of life
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard physical therapy program (Sham Comparator): all participants will receive strengthing, stretching, facilitation and inhibitory techniques, splinting, developmental techniques, gait, and balance training. The duration of each session will be 1 hour, 3 times per week for 4 weeks.
  Interventions: Other: Standard physical therapy program
- Radial shockwave therapy (rSWT) (Active Comparator): One session per week of rSWT will be applied using shockwave device. The following parameters will be used: Shocks number: 1500 per muscle, will be applied over the belly of the calf muscle using the 15 mm applicator head. The pressure will be 2 bar and the frequency will be 4 Hz. Patients will receive shock wave from prone position.
  Interventions: Other: Experimental Interventions

INTERVENTIONS:
Other: Experimental Interventions — One session per week of rSWT will be applied using the BMI-1120 SHOCK MED device (BIO-MED-INC- ITALY). The following parameters will be used: Shocks number: 1500 per muscle, will be applied over the belly of the calf muscle using the 15 mm applicator head. The pressure will be 2 bar and the frequency will be 4 Hz. Patients will receive shock wave from prone position.
  Other Names: Radial shock wave therapy (rSWT)
  Arms: Radial shockwave therapy (rSWT)
Other: Standard physical therapy program — Regular rehabilitation procedures consist of strengthing, stretching, facilitation and inhibitory techniques, splinting, developmental techniques, gait and balance training, and advice to parents. The duration of each session will be 1 hour, 3 times per week for 4 weeks
  Other Names: Standard physical therapy intervention
  Arms: Standard physical therapy program

SUMMARY:
the aim of this study to assess different outcome measures after applying standard physical therapy plus radial shockwave and compare the results with another group who received standard treatment only.

Design: double-blinded (assessor and data analyzer)

Methods: This study will be conducted in 4 rehabilitation facilities, Times for 1 month of intervention Assessment timeline: 3 times (T0: at baseline, T1: at 4 weeks, T2: follow up at 3 months. Outcome measures: the Modified Ashworth scale (MAS), Ankle ROM, Plantar surface area, Gross motor function, and quality of life

DETAILED DESCRIPTION:
the current study is a randomized controlled trial in which the researchers intended to examine the effect of adding radial shockwave therapy to standard physical therapy on the status of calf muscle spasticity and consequent effects on gross motor function, ankle joint ROM, plantar surface area, and quality of life.

the experimental intervention will consist of 4 sessions of radial shockwave applied to the bulkiest area of the calf muscle in children having spastic cerebral palsy. participants will receive 1 session of radial shockwave per week and will continue their regular physical therapy as usual (3 sessions per week).

outcome assessment will be conducted 3 times: at baseline, after the end of the treatment program, and at 3 months follow-up.

the tools that will be used to collect data will be:

1. Modified Ashworth scale for muscle tone.
2. Goniometer for Ankle ROM.
3. EMed force platform for plantar surface area
4. Gross motor function scale for gross motor function
5. Cerebral Palsy Quality of Life Questionnaire for quality of life assessment

ELIGIBILITY:
Inclusion Criteria:

* age between 8-14
* diagnosed with spastic CP
* ability to walk alone or with assistance
* grades 1 -4 on Gross Motor Function Classification System
* at least score 1 on the Modified Ashworth Scale (MAS)
* ability to attend the treatment program and the outcome assessment sessions.

Exclusion Criteria:

* patients who received a botulinum toxin injection in the calf muscle during the last six months
* structural contracture of the calf muscle
* surgery in the lower extremity during the previous year
* those experiencing pain in the lower limbs
* severe associated neurological diseases as epilepsy
* medications affecting peripheral muscle tone.

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2024-02-13 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
calf muscle tone | at baseline
  the Modified Ashworth scale (MAS) will be used to assess the tone of the affected calf muscle. the test will be done by moving the ankle joint passively and assess quality of movement and resistance provided by the tissues. scores ranged from 0 to 4 where 0 means normal and 4 means higher spasticity
calf muscle tone | at 4 weeks
  the Modified Ashworth scale (MAS) will be used to assess the tone of the affected calf muscle. the test will be done by moving the ankle joint passively and assess quality of movement and resistance provided by the tissues. scores ranged from 0 to 4 where 0 means normal and 4 means higher spasticity
calf muscle tone | at follow up (3months after the end of the treatment)
  the Modified Ashworth scale (MAS) will be used to assess the tone of the affected calf muscle. the test will be done by moving the ankle joint passively and assess quality of movement and resistance provided by the tissues. scores ranged from 0 to 4 where 0 means normal and 4 means higher spasticity
ankle joint ROM | at baseline
  traditional goniometer will be used to measure active ROM of the ankle joint. the patient will be in supine position during assessment
ankle joint ROM | at 4 weeks
  traditional goniometer will be used to measure active ROM of the ankle joint. the patient will be in supine position during assessment
ankle joint ROM | at follow up (3months after the end of the treatment)
  traditional goniometer will be used to measure active ROM of the ankle joint. the patient will be in supine position during assessment
plantar surface area | at baseline
  E Med force platform will be used to assess plantar surface area during normal relaxed standing. it will be expected that larger surface area indicate improvement in calf muscle spasticity
plantar surface area | at 4 weeks
  E Med force platform will be used to assess plantar surface area during normal relaxed standing. it will be expected that larger surface area indicate improvement in calf muscle spasticity
plantar surface area | at follow up (3months after the end of the treatment)
  E Med force platform will be used to assess plantar surface area during normal relaxed standing. it will be expected that larger surface area indicate improvement in calf muscle spasticity
gross-motor function | at baseline
  Gross Motor Function Measure scale will be used to assess changes in gross motor. function in cerebral palsy patients. the score will be determined according to the tasks the patient can do. where lower score (1) for nealy normal patients while score of (5) will indicate lowest gross motor abilities.
gross-motor function | at 4 weeks
  Gross Motor Function Measure scale will be used to assess changes in gross motor. function in cerebral palsy patients. the score will be determined according to the tasks the patient can do. where lower score (1) for nealy normal patients while score of (5) will indicate lowest gross motor abilities.
gross-motor function | at follow up (3months after the end of the treatment)
  Gross Motor Function Measure scale will be used to assess changes in gross motor. function in cerebral palsy patients. the score will be determined according to the tasks the patient can do. where lower score (1) for nealy normal patients while score of (5) will indicate lowest gross motor abilities.

SECONDARY OUTCOMES:
cerebral palsy quality of life questionnaire | at baseline
  Parents will be asked to report their level of quality of life using the Cerebral Palsy Qualityof life questionnair. the higher the gained score the better the quality of life achieved.
cerebral palsy quality of life questionnaire | at 4 weeks
  Parents will be asked to report their level of quality of life using the Cerebral Palsy Qualityof life questionnair. the higher the gained score the better the quality of life achieved.
cerebral palsy quality of life questionnaire | at follow up (3months after the end of the treatment)
  Parents will be asked to report their level of quality of life using the Cerebral Palsy Qualityof life questionnair. the higher the gained score the better the quality of life achieved.

CONTACTS AND LOCATIONS:
Overall Officials: Hisham M Hussein, PHD, Principal Investigator — University of Hail
Locations (1):
- King Salman Hospital, Hail, Saudi Arabia